CLINICAL TRIAL: NCT02291770
Title: Treatment of of Chronic Graft-Versus-Host Disease With Mesenchymal Stromal Cells. A Phase III Randomized Open Label Multi-center Study in Southern China.
Brief Title: Treatment of Chronic Graft-Versus-Host Disease With Mesenchymal Stromal Cells
Acronym: MSC-cGvHD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Sun Yat-sen University (Other); Nanfang Hospital, Southern Medical University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Academy Military Medical Science, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.GRDEC 2014210H
Record Dates: First submitted 2014-11-05; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Graft-Versus-Host Disease
Keywords: Chronic Graft-Versus-Host Disease; Mesenchymal Stromal Cells
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cells (MSC) (Active Comparator): Patients with newly diagnosed cGvHD receive primary treatment plus MSC:
  1. MSC+prednisone+cyclosporine;
  2. MSC+prednisone+tacrolimus;
  3. MSC+prednisone+mycophenolate mofetil.
  Interventions: Biological: Mesenchymal Stromal Cells
- Placebo (Placebo Comparator): Patients with newly diagnosed cGvHD receive primary treatment:
  1. Placebo+prednisone+cyclosporine;
  2. Placebo+prednisone+tacrolimus;
  3. Placebo+prednisone+mycophenolate mofetil.

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells — Mesenchymal stem cell(MSC). Patients with newly diagnosed cGvHD: prednisone 1mg/kg + cyclosporine or tacrolimus and MSC 2×1,000,000 MSC/kg, IV twice a week for the first two weeks and weekly for the following two weeks(6 doses totally).
  Other Names: MSC
  Arms: Mesenchymal stem cells (MSC)

SUMMARY:
Chronic Graft-versus-Host Disease (cGvHD) is a potentially lethal disorder. A variety of second line immunosuppressive agents have been investigated but no optimal treatment has emerged. There is therefore a need for novel treatment strategies. Mesenchymal stromal cells (MSC) exhibit immunomodulatory properties and a recent pilot study suggests a response rate of 70% in steroid- refractory patients. In the present randomized study the efficacy and safety of MSC treatment will be further studied in patients with cGvHD.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cGvHD
* Informed consent obtained from patient and donor.
* Any patient who has undergone allogeneic stem cell transplantation with c GvHD.
* Have not received additional agent for cGVHD within 3 months.
* Expected life is more than 90 days.
* Adequate pulmonary function with no evidence of chronic obstructive or severe restrictive pulmonary disease.
* Adequate cardiac function with no evidence of uncontrolled high blood pressure,congestive heart failure, angina pectoris, acute myocardial infarction within 6 months prior to the process.

Exclusion Criteria:

* Invasive fungal disease.
* Active cytomegalovirus (CMV)/Epstein-Barr virus(EBV)/varicella disease).
* Patient is with a history of hypersensitivity to bovine products.
* Relapsed malignancy.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients responding to treatment of cGvHD with MSC | 90 days

SECONDARY OUTCOMES:
Overall survival | 2 year
Progression-free survival | 2 year
Time without systemic immunosuppression | 2 year
Cumulative incidents of non-relapse mortality | 2 year
Adverse events | 2 year

OTHER OUTCOMES:
Quality of life | 2 year
Immune reconstitution including monitoring of absolute T-cell subsets, B-cells, NK-cells as well as biomarkers of cGvHD | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Xin Du, Prof., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Xin Du, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Weng J, He C, Lai P, Luo C, Guo R, Wu S, Geng S, Xiangpeng A, Liu X, Du X. Mesenchymal stromal cells treatment attenuates dry eye in patients with chronic graft-versus-host disease. Mol Ther. 2012 Dec;20(12):2347-54. doi: 10.1038/mt.2012.208. Epub 2012 Oct 16. PMID 23070118
- [Background] Weng JY, Du X, Geng SX, Peng YW, Wang Z, Lu ZS, Wu SJ, Luo CW, Guo R, Ling W, Deng CX, Liao PJ, Xiang AP. Mesenchymal stem cell as salvage treatment for refractory chronic GVHD. Bone Marrow Transplant. 2010 Dec;45(12):1732-40. doi: 10.1038/bmt.2010.195. Epub 2010 Sep 6. PMID 20818445